CLINICAL TRIAL: NCT07275918
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SA1211 Injection in Healthy Participants and Participants With Chronic Hepatitis B
Brief Title: SA1211 Injection Phase 1 Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Siran Biotechnology Co.,Ltd. (Industry)
Collaborators: Beijing Siran Biotechnology Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHB101
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis B
Keywords: CHB
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Experimental)
  Interventions: Drug: SA1211 injection; Drug: SA1211 injection placebo
- Chronic Hepatitis B (Experimental)
  Interventions: Drug: SA1211 injection; Drug: SA1211 injection placebo

INTERVENTIONS:
Drug: SA1211 injection — subcutaneous injection
Drug: SA1211 injection placebo — subcutaneous injection

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, immunogenicity and Pharmacokinetics (PK) characteristics of SA1211 Injection in healthy volunteers (Part A) and participants with chronic hepatitis B (CHB, Part B), and assess its preliminary efficacy in participants with chronic hepatitis B (CHB). The main questions it aims to answer are:

What are the safety, tolerability, immunogenicity and PK characteristics of a single subcutaneous injection of SA1211 Injection in healthy volunteers (Part A)? What are the safety, tolerability, immunogenicity and PK characteristics of multiple subcutaneous injections of SA1211 Injection in participants with CHB (Part B)? What is the preliminary efficacy of SA1211 Injection in participants with CHB (Part B)?

Participants will:

* Part A (healthy volunteers): Receive a single subcutaneous injection of SA1211 Injection or placebo and complete relevant safety, tolerability and PK monitoring as required.
* Part B (participants with CHB): Receive multiple subcutaneous injections of SA1211 Injection or placebo and complete relevant safety, tolerability, PK monitoring and preliminary efficacy assessment as required.

ELIGIBILITY:
Inclusion Criteria:

1. Able to correctly understand and sign the informed consent form in writing.
2. Male or female participants.

   * For healthy participants: aged 18-55 years old (inclusive of the cut-off values).
   * For participants with chronic hepatitis B (CHB): aged 18-65 years old (inclusive of the cut-off values).
3. Body Mass Index (BMI) meets the following requirements.

   * For healthy participants: within the range of 18-28 kg/m² (inclusive of the cut-off values).
   * For participants with chronic hepatitis B (CHB): within the range of 18-32 kg/m² (inclusive of the cut-off values).
4. During the screening period, the results of the following examinations are either normal or abnormal but not clinically insignificant:

   - Clinical laboratory tests: complete blood count, blood biochemistry, coagulation function, urine routine. Thyroid function test. 12-lead electrocardiogram (ECG). Abdominal ultrasound. Posteroanterior chest X-ray.
5. For participants with chronic hepatitis B (CHB): documented hepatitis B virus (HBV) infection for at least 6 months before screening, with positive hepatitis B surface antigen (HBsAg) and/or positive HBV deoxyribonucleic acid (HBV DNA).
6. For female participants of childbearing potential: must not be pregnant or lactating, and agree to use effective contraception during the study period.
7. For male participants of childbearing potential: agree to use effective contraception during the study period to ensure effective contraception for their sexual partners.

Exclusion Criteria:

1. Participants with concurrent hepatitis C virus (HCV), human immunodeficiency virus (HIV) or syphilis infection; or those previously diagnosed with hepatitis A, D, or E who have not been cured.
2. Participants with severe diseases, including but not limited to diseases of the nervous, cardiovascular, hematological and lymphatic, immune, renal, hepatic, thyroid, gastrointestinal, respiratory, metabolic, and skeletal systems, as well as a history of malignant tumors.
3. Participants with severe mental illness or uncontrolled mental disorders, including but not limited to schizophrenia, bipolar disorder, or depression.
4. Participants with a systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at screening, who are deemed unsuitable for the study by the investigator.
5. Participants who have undergone major surgery within 6 months before screening, or plan to undergo surgery during the study period.
6. Participants with severe infection or trauma within 4 weeks before screening.
7. Participants with a severe allergic constitution, or a confirmed allergy to this product or its formulation components.
8. Participants who smoked more than 5 cigarettes per day or the equivalent amount of tobacco within 3 months before screening.
9. Participants deemed unsuitable for the trial by the investigator due to other factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AEs, SAEs and abnormal laboratory testings | Approximate 24 weeks
  AEs: Adverse Events. SAEs: Serious Adverse Events.

SECONDARY OUTCOMES:
Cmax: maximum concentration | Pre-dose, multiple time-points post dose until 48 hours
Tmax | Pre-dose, multiple time-points post dose until 48 hours
  Tmax: Time to Maximum Concentration
AUC0-t | Pre-dose, multiple time-points post dose until 48 hours
  AUC0-t: Area Under the Concentration-Time Curve from Time Zero to the Last Quantifiable Concentration
AUC0-inf | Pre-dose, multiple time-points post dose until 48 hours
  AUC0-inf: Area Under the Concentration-Time Curve from Time Zero to Infinity
t1/2 | Pre-dose, multiple time-points post dose until 48 hours
  t1/2: Half-life
λz | Pre-dose, multiple time-points post dose until 48 hours
  λz: Terminal Elimination Rate Constant
Vd/F | Pre-dose, multiple time-points post dose until 48 hours
  Vd/F: Volume of Distribution over Bioavailability
CL/F | Pre-dose, multiple time-points post dose until 48 hours
  CL/F: Clearance over Bioavailability
Css (Steady-State Concentration) | Pre-dose, multiple time-points post dose until 48 hours
DF (Degree of Fluctuation) | Pre-dose, multiple time-points post dose until 48 hours
The number of participants with chronic hepatitis B (CHB) who achieved hepatitis B surface antigen (HBsAg) clearance | Approximate 24 weeks
Maximum HBsAg Decline in CHB Participants Within 24 Weeks (log10) | Approximate 24 weeks
The number of CHB Participants with HBsAg Seroconversion at each assessment time Point within 24 weeks | Approximate 24 weeks
The number of CHB participants who achieved HBeAg seronegativity at each assessment time point within 24 weeks | Approximate 24 weeks
The number of participants with immunogenicity (i.e., anti-drug antibodies [ADAs]) | Approximate 24 weeks
The change in QTcF relative to baseline and the change relative to placebo | Approximate 24 weeks
  Apply for healthy participants

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No